CLINICAL TRIAL: NCT00640367
Title: Synthesis Expansion: A Randomized Controlled Trial on Intra-Arterial Versus Intravenous Thrombolysis in Acute Ischemic Stroke
Brief Title: Intra-arterial Versus Systemic Thrombolysis for Acute Ischemic Stroke
Acronym: SYNTHESIS EXP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYNTHESIS EXPANSION
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: Acute ischemic stroke; thrombolysis; intra-arterial thrombolysis
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IA thrombolysis (Experimental): IA recombinant tissue plasminogen activator and/or mechanical thrombolysis
  Interventions: Other: Alteplase IA and/or mechanical thrombolysis
- IV rtPA (Active Comparator): IV recombinant tissue plasminogen activator
  Interventions: Drug: Alteplase IV

INTERVENTIONS:
Other: Alteplase IA and/or mechanical thrombolysis — loca intra-arterial recombinant tissue plasminogen activator and/or mechanical thrombolysis
  Arms: IA thrombolysis
Drug: Alteplase IV — intravenous recombinant tissue plasminogen activator
  Arms: IV rtPA

SUMMARY:
SYNTHESIS is a pragmatic multicenter randomized controlled trial (RCT), open-label, with blinded follow-up aiming to determine whether loco-regional intra-arterial (IA) with recombinant tissue-plasminogen activator (rt-PA) and/or mechanical devices, as compared with systemic intravenous (I.V.) infusion of rt-PA within 3 hours of ischemic stroke, increases the proportion of independent survivors at 3 months.

DETAILED DESCRIPTION:
Eligibility criteria:patients with symptomatic, CT verified, acute ischemic stroke, being able to initiate IV rt-PA within 3 hours and IA thrombolysis within 6 hours of stroke onset, when uncertainty about appropriateness the two approaches exists as established by the treating physician.

Eligible patients are randomized to receive either 0.9 mg/kg (max 90 mg) IV rt-PA (control arm) or up to 0.9 mg/Kg IA rt-PA (max 90 mg) over 60 minutes into the thrombus, eventually associated with clot mechanical disaggregation/dislocation or retraction/aspiration. Mechanical thrombolysis is possible also without the use of rt-PA. The procedural choices of the interventional neuroradiologist depend on the type of occlusion, circumstances and experience.

The study is designed to detect or disprove (alpha=5% and power probability=80%) a 15% absolute difference between the treatment groups in the percentage of patients with a favourable outcome (Modified Rankin Scale Score = 0-1).Enrollment will be completed with 350 randomized patients.

Neurological deficit will be scored with NIH Stroke Scale at day 7 or discharge, or transfer to another hospital, whichever occurs first.Patient's clinical condition will be again evaluated by a telephone call after 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Sudden focal neurological deficit attributable to a stroke
* Clearly defined time of onset, allowing initiation of intravenous treatment within 3 hours of symptoms onset and intra-arterial treatment within 6 hour of symptoms onset.
* Age greater than 18 years

Exclusion Criteria:

* Disability preceding stroke consistent with a modified Rankin scale score of 2-4
* Coma at onset
* Rapidly improving neurological deficit
* Seizure at onset
* Clinical presentation suggestive of a subarachnoid hemorrhage
* Previous history of intracranial hemorrhage
* Septic embolism
* Arterial puncture at a non compressible site within the previous 7 days
* Any traumatic brain injury within the previous 14 days
* Surgery of the central nervous system in the previous 3 months
* Gastrointestinal hemorrhage or urinary tract hemorrhage within the previous 14 days.
* Current therapy with intravenous or subcutaneous heparin to rise the clotting time
* Known hereditary or acquired hemorrhagic diathesis, baseline INR greater than 1.5, aPTT more than 1.5 times normal, or baseline platelet count less than 100,000 per cubic millimeter
* Baseline blood glucose concentrations below 2.75 mm/L (50 mg/dL).
* Known contrast sensitivity.
* Women of childbearing potential (unless pregnancy impossible) or known to be breastfeeding. Uncontrolled hypertension defined by a blood pressure greater or equal 185 mmHg systolic or diastolic greater or equal 110 mm Hg in 3 separate occasions at least 10 minutes apart or requiring continuous IV therapy.
* Prognosis very poor regardless of therapy; likely to be dead within months.
* Unlikely to be available for follow-up (eg, no fixed home address, visitor from overseas).
* Any other condition which local investigators feels would pose a significant hazard in terms of risk/benefit to the patient, or if therapies are impracticable.

COMPUTED TOMOGRAPHIC (CT) SCAN EXCLUSION CRITERIA

* Intracranial tumors except small meningioma
* Hemorrhage of any degree
* Acute infarction (since this may be an indicator that the time of onset is uncorrected)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To assess whether IA thrombolysis, as compared to IV rt-PA, increases survival free of disability (modified Rankin score of zero or 1) at 3 months. | 3 months

SECONDARY OUTCOMES:
To asses whether IA thrombolysis vs.IV rt-PA 1.improves the 7 day neurological deficit; 2.is safe on the base of symptomatic intracranial hemorrhages, fatal and non-fatal stroke, death from any cause, neurological deterioration within 7 days | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Ciccone, MD, Principal Investigator — A.O. Ospedale Niguarda Ca' Granda
Locations (1):
- A.O. Ospedale Ca' Granda, Milan, Milan, Italy

REFERENCES:
- [Derived] Ciccone A, Valvassori L, Nichelatti M, Sgoifo A, Ponzio M, Sterzi R, Boccardi E; SYNTHESIS Expansion Investigators. Endovascular treatment for acute ischemic stroke. N Engl J Med. 2013 Mar 7;368(10):904-13. doi: 10.1056/NEJMoa1213701. Epub 2013 Feb 6. PMID 23387822